CLINICAL TRIAL: NCT02242812
Title: Telmisartan Effectiveness on Left Ventricular MAss Reduction (TELMAR) as Assessed by MRI, in Patients With Mild to Moderate Hypertension - a Prospective, Randomised, Double-blind Comparison of Telmisartan 80 mg Oral, Once Daily, to Metoprolol Succinate 95 mg Oral, Once Daily, Over a Period of 6 Months
Brief Title: Telmisartan Effectiveness on Left Ventricular Mass Reduction (TELMAR) as Assessed by MRI, in Patients With Mild to Moderate Hypertension
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 502.393
Record Dates: First submitted 2014-09-16; First posted 2014-09-17 (Estimated); Last update posted 2014-09-17 (Estimated); Status verified 2014-09

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Telmisartan; Metoprolol

ARMS (2):
- Telmisartan (Experimental): MICARDIS®
  Interventions: Drug: Telmisartan; Drug: Placebo
- Metoprolol succinate (Active Comparator): BELOC ZOK®
  Interventions: Drug: Metoprolol succinate; Drug: Placebo

INTERVENTIONS:
Drug: Telmisartan
  Arms: Telmisartan
Drug: Metoprolol succinate
  Arms: Metoprolol succinate
Drug: Placebo

SUMMARY:
The primary objective was to show that telmisartan is not inferior to metoprolol succinate in respect of the percentage change from baseline in LVMI(H) after a 6.5 months treatment period. As secondary objectives, the improvement in left ventricular systolic and diastolic function and blood pressure reduction were assessed

ELIGIBILITY:
Inclusion Criteria:

* Caucasian and non-Caucasian patients i.e. Asian patients with untreated essential hypertension as defined by either a mean systolic blood pressure (SBP) of >= 140 mm Hg or a mean diastolic blood pressure (DBP) of >= 90 mm Hg during normal daily activities (6:00 - 21:59 h) and/or a nocturnal (22:00 - 05:59 h) SBP mean of >= 120 mm Hg or a DBP mean of >= 70 mm Hg as measured by ABPM.
* Presence of Left Ventricular Hypertrophy (LVH) as defined by MRI:

  * Caucasian patients: Left ventricular mass of > 0.8 g/cm for women or > 1.05 g/cm for men. Non-Caucasian i.e. Asian patients: Left ventricular mass of > 0.65 g/cm for women or > 0.85 g/cm for men
* Age between 18 and 80 years
* Written informed consent in accordance with Good Clinical Practice (GCP) guidelines and the local regulatory and legal requirements

Exclusion Criteria:

* Contraindications to the class of drugs under study:

  * Contraindications against β Blocker or angiotensin receptor antagonists
  * A history of angioedema or known hypersensitivity to any component of the formulations
* Contraindications on ethical grounds:

  * there are no specific contraindications ethical grounds foreseen in this study
* General Contraindications:

  * Pregnancy, lactation or child bearing potential (I.e. Pre-menopausal women (last menstruation < 1 year prior to start of run-in phase) who are not surgically sterile (hysterectomy, tubal ligation) or who are NOR practicing or do NOT plan to practice acceptable means of birth control (Intrauterine Device, oral implantable or injectable contraceptives) or who have a positive serum pregnancy test at screening or baseline)
  * Factors making follow up difficult (i.e. no fixed address)
  * Treatment with other investigational drugs within one month of signing informed consent
* Clinically significant concomitant diseases:

  * Hepatic and/or renal dysfunction as defined by the following laboratory parameters:

    1. Alanine amino transferase (SGPT (ALT)) or Aspartate amino transferase (SGOT (AST)) values above two times or Gamma glutaryl transferase (Gamma-GT) three times the upper normal limit
    2. Serum creatinine > 150 mol/L
  * Clinically significant sodium or potassium depletion, clinically relevant hyperkalaemia
  * Uncorrected volume depletion
  * Primary aldosteronism
  * Hereditary fructose intolerance
  * Biliary obstructive disorders, cholestasis or moderate to severe hepatic insufficiency
  * Insulin-dependent diabetes mellitus
  * Congestive heart failure or ejection fraction < 35% New York Heart Association (NYHA) class III or IV
  * Unstable Angina
  * Sustained ventricular tachycardia, atrial fibrillation, atrial flutter or other clinically relevant cardiac arrhythmias as determined by the investigator
  * Post-renal transplant patients
  * Myocardial infarction or cardiac surgery within the preceding six months
* Known drug or alcohol abuse within 6 months prior to start of study
* Patients with MRI contraindications:

  * Implanted pacemaker or defibrillator
  * Implanted vascular clips
  * Gross obesity (i.e. patients weight > 150 kg)
* Specific exclusion for the disease under study:

  * Known or suspected secondary hypertension
  * Known renal artery stenosis
  * Known endocrine disorders with secondary hypertension
  * Severe arterial hypertension as defined by a mean seated DBP > 115 mmHg or a mean seated SBP > 200 mmHg
  * Patients with a complete loss of diurnal BP variation, as defined by the lack of drop of BP during sleeping time or a drop of less than 5% when compared to daily mean BP
  * Hypertrophic obstructive cardiomyopathy, clinically relevant aortic valve stenosis or clinically relevant mitral valve disease; vascular disease affecting BP (coarctation; stenosis of A. subclavia)
* Specific concomitant therapy exclusions:

  * Use of antihypertensive medication within the previous six months
  * Chronic administration of digoxin or other digitalis-type drugs, without regular monitoring of plasma level
  * Chronic administration of any medications known to affect blood pressure, except medications allowed by the protocol
  * Continuous (for more than two weeks) treatment within the last three months using at least on of the following drugs: β blockers, angiotensin converting enzyme inhibitors, angiotensin receptor blockers
* Participation in another drug trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2003-09; Primary Completion 2004-10 (Actual)

PRIMARY OUTCOMES:
Percentage change in left ventricular mass index relative to height (LVMI(H)) | Baseline, day 180
  based on LVM measurements by magnetic resonance imaging (MRI)

SECONDARY OUTCOMES:
Number of patients with adverse events | up to 6.5 months
Change of left ventricular mass index related to the body surface area (LVMI (BSA)) measured by MRI | Baseline, day 180
Change of left ventricular end-systolic (LVESV) measured by MRI | Baseline, day 180
Change of left ventricular end-diastolic volume (LVEDV) as measured by MRI | Baseline, day 180
Change of left ventricular end-diastolic volume index related to height LVEDVI (H)) | Baseline, day 180
  based on LV volumetric measurements by MRI
Change of left ventricular end-diastolic volume index related to the body mass index (LVEDVI (BSA)) | Baseline, day 180
  based on LV volumetric measurements by MRI
Change of left ventricular ejection fraction (EF) | Baseline, day 180
  based on LV volumetric measurements by MRI
Change of end-systolic wall stress (ESWS) measured by MRI | Baseline, day 180
Change of 24-hour mean systolic blood pressure measured by ambulatory blood pressure monitoring (ABPM) | Baseline, day 179
Change of 24-hour mean diastolic blood pressure as measure by ABPM | Baseline, day 179
Change of mean seated trough systolic blood pressure measured by manual cuff sphygmomanometer | up to day 194
Change of mean seated trough diastolic blood pressure measured by manual cuff sphygmomanometer | up to day 194